CLINICAL TRIAL: NCT03769740
Title: Cerebral Oximetry and NIRS in Cardiac Arrest Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Brian O'Neil, Professor and Chair of Department of Emergency Medicine, Wayne State University
Other Study IDs: 047609MP4E
Record Dates: First submitted 2018-11-08; First posted 2018-12-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Death; Cardiac Arrest; Emergencies
Keywords: cardiac arrest, cardiac death, CPR, neurologic prognostication, emergency medicine,
MeSH Terms: conditions — Death; Heart Arrest; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- CPR Group
  Interventions: Device: Cerebral Oximetry

INTERVENTIONS:
Device: Cerebral Oximetry — Non invasive, near infrared spectroscopy cerebral oximetry

SUMMARY:
This is an observational study to define the role and future applications of cerebral oximetry in cardiac arrest patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Non-traumatic cardiac arrest or post non-traumatic cardiac arrest
* No purposeful response to verbal or noxious stimuli

Exclusion Criteria:

* Age < 18 years
* Open head injury/trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department experiencing non-traumatic cardiac arrest or arriving post non-traumatic cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
ROSC | During ED resuscitation
  Return of spontaneous circulation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - DMC Detroit Receiving Hospital - Wayne State University, Detroit, Michigan
  - DMC Sinai-Grace Hospital, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Undecided